CLINICAL TRIAL: NCT03546673
Title: Expressive Writing Among Chinese Breast Cancer Survivors: Study One
Brief Title: Health Benefits of Expressive Writing: Study One
Acronym: Komen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Herald Cancer Association (Other); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Qian Lu, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 09021-02
Record Dates: First submitted 2018-05-18; First posted 2018-06-06 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Chinese breast cancer survivors expressive writing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Condition (No Intervention): Participants in the control group were asked to write for three weeks about facts regarding their cancer and its treatment for three sessions.
- Self-regulation Condition (Experimental): For the self-regulation condition, each weekly writing assignment covers a different task. During session one, participants will be asked to write about their deepest feelings and thoughts regarding their experience with breast cancer as well as its impact on their lives; in session two, participants will be asked to write about their coping strategies to deal with stressors associated with the cancer diagnosis and treatment, as well as future plans for coping with cancer-related stressors; and in session three, participants will be asked to write about positive thoughts and feelings regarding their experience with breast cancer.
  Interventions: Behavioral: Self-Regulation Condition
- Emotional Disclosure condition (Experimental): For the emotional disclosure condition, participants were asked to write about their deepest thoughts and feelings about their cancer experience for three weeks.
  Interventions: Behavioral: Emotional Disclosure Condition

INTERVENTIONS:
Behavioral: Self-Regulation Condition
  Arms: Self-regulation Condition
Behavioral: Emotional Disclosure Condition
  Arms: Emotional Disclosure condition

SUMMARY:
This study is a randomized controlled trial (RCT) with the aim of determining the cultural sensitivity, feasibility, and effectiveness of an expressive writing intervention for Chinese breast cancer survivors.

DETAILED DESCRIPTION:
The study examines the potential health benefits (i.e., physical health, psychological health, and quality of life) of this expressive writing intervention for Chinese-speaking breast cancer survivors. The study also explores the mechanism through which expressive writing confers health benefits and investigates who will benefit most from the expressive writing intervention. Chinese-speaking breast cancer survivors who have completed primary treatment will be randomly assigned to a control writing condition, a self-regulation condition, or an emotional disclosure writing condition. Health outcomes are assessed at baseline, and 1, 3, and 6 months follow-ups. Mixed qualitative-quantitative mixed methods are used to explore the effect of the intervention on health outcomes and explore the mechanisms that explain the benefits of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* 1) having a breast cancer diagnosis
* 2) completing primary medical treatment within four years
* 3) being comfortable writing and speaking Chinese (i.e. Mandarin or Cantonese)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in quality of life score as assessed by Functional Assessment of Cancer Therapy Scale (FACT). | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The Functional Assessment of Cancer Therapy Scale (FACT) is a 27-item measure of health-related quality of life (Cella & Tulsky,1993), which assesses perceived life quality in four different facets, including physical well-being (7 items), social well-being (7 items), emotional well-being (6 items), and functional wellbeing (7 items).

SECONDARY OUTCOMES:
Change in Post-traumatic stress symptoms assessed by The PTSD Symptom Scale - Self Report | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 17 items reflecting the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition -Text Revision (DSM-IV-TR) symptoms of post-traumatic stress disorder (Foa, Riggs, Dancu, & Rothbaum, 1993).
Change in fatigue as assessed by Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The FACIT-F scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week (Webster et al., 2003).
Change in perceived pain assessed by Brief Pain Inventory short form. | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The Brief Pain Inventory-short form is a 9-item inventory which assesses the severity of pain and its impact on functioning (Cleeland, 1991).
Change in sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989).
Change in physical symptoms as assessed by the Physical Symptoms Checklist | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The 10-item symptom questionnaire was used to assess the number of days during the last 30 days which participants had felt symptoms of acute illness such as runny nose, difficulty in breathing and soreness during the past month not due to intentional physical exercise.This measure was modified from Pennebaker (1982) and King and Emmons (1990).

OTHER OUTCOMES:
Change in positive and negative affect assessed by the Positive and negative affect scale | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 20 items that measure positive and negative affect (Watson, Clark, & Tellegen, 1988).
Change in fear of cancer recurrence assessed by one item statement "I worry that my cancer will come back" | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  On the statement "I worry that my cancer will come back", participants rate their agreement with this statement on a 5-point scale from "not at all" to "very".
Change in cancer-related morbidity | Immediately after the intervention through 3 months after the intervention
  Patients will prospectively record all medical visits during the period from the end of intervention through the subsequent 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, Ph.D., MD, Principal Investigator — University of Houston
Locations (2):
- United States (2):
  - Herald Cancer Association, Los Angeles, California
  - University of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu Q, Wong CCY, Lu Q. Acculturation Moderates the Effects of Expressive Writing on Post-Traumatic Stress Symptoms Among Chinese American Breast Cancer Survivors. Int J Behav Med. 2019 Apr;26(2):185-194. doi: 10.1007/s12529-019-09769-4. PMID 30656609